CLINICAL TRIAL: NCT04552249
Title: Evaluation of Age-related Skin Changes and Instrument Reliability Using Clinical Probe Measurements and Imaging Modalities
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-604-000
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Age-related Skin Changes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1
- Group 2
- Group 3
- Group 4
- Group 5
- Group 6

SUMMARY:
To evaluate the reliability of different non-invasive skin probe measurements.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type I to VI with about 15% of phototypes V/VI.
* Subject agreeing to complete all study required procedures.
* Subject having given freely and expressly his/her informed consent.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment.
* Subject participating to another research on human beings or being in an exclusion period for a previous study.
* Intensive exposure to sunlight or UV-rays within the previous month and foreseen during the study.
* Subject who underwent tissue augmentation with dermal fillers including HA, calcium hydroxylapatite, autologous fat, mesotherapy, or other cosmetic procedures (eg, face-lift, laser, photomodulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, or other ablative procedures) in the face within 12 months before study entry or was planning to undergo any such treatment during the study.
* Subject who underwent treatment with botulinum toxins in the face or neck within 6 months of study entry or was planning to undergo such treatment during the study.
* Subject who ever received semi-permanent fillers or permanent facial implants (eg, poly-L-lactic acid, polymethylmethacrylate, silicone, expanded polytetrafluoroethylene) anywhere in the face or was planning to be implanted with any of these products at any time during the study.
* Subject with current cutaneous inflammatory or infectious processes (eg, acne, herpes), abscess, an unhealed wound, or a cancerous or precancerous lesion on the face that could interfere with measurements.
* Subject having changed, started or stopped any hormonal treatment or any treatment likely to have an impact on skin condition (over-the-counter or prescription, oral or topical, anti-wrinkle products on the face), within 30 days prior to enrollment or is planning to begin using such products during the study.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 subjects will be included, with at least 25 subjects per group
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Age-related changes in skin hydration on the cheek | 2 Months
  Skin hydration will be measured using tissue dielectric constant measurement. Tissue dielectric constant is expressed as a unitless value that is directly proportional to the amount of water in the tissue.
Age-related changes in skin elasticity on the cheek | 2 Months
  Skin elasticity measurement using suction based device
Age-related changes in skin color on the cheek | 2 Months
  Skin colorimetric measurement will be done with a Spectrophotometer
Age-related changes in skin thickness on the cheek | 2 Months
  Epidermal thickness will be measured with an optical coherence tomography instrument
Age-related changes in skin blood flow on the cheek | 2 Months
  Blood Flow (redness) will be measured with an optical coherence tomography instrument
Age-related changes in skin roughness on the cheek | 2 Months
  Skin surface roughness will be measured with an optical coherence tomography instrument
Age-related changes in skin OAC on the cheek | 2 Months
  Optical Attenuation Coefficient (OAC) will be measured with an optical coherence tomography instrument
Age-related changes in skin topography on the cheek | 2 Months
  Skin topography imaged using a using a fringe projection imaging system. Output measurements from the images will include Ra (average roughness), Rq (Root Mean Square of the profile heights), RMax (Maximum Roughness Depth), Rv (Depth of the Largest Profile Valley), Rvm (Average depth of the Profile Valleys), Rz (average height of roughness) and Rt (maximum height of the roughness profile).
Age-related changes in skin gloss on the cheek | 2 Months
  Skin gloss (Shine and Oiliness) imaged using a camera-based system which uses various lighting/capture modalities to enhance the visualization of skin features
Age-related changes in fine lines on the cheek | 2 Months
  The investigator will assess the participant's appearance of fine lines/wrinkles using a 5-point scale from (0=None to 4=Diffuse)
Clinical scoring of age-related changes in skin roughness on the cheek | 2 Months
  The investigator will assess the participant's appearance of skin roughness using a 5-point scale from (0=None to 4=Diffuse)

SECONDARY OUTCOMES:
To evaluate the reliability of skin hydration measurement on the cheek between different time points and different technicians. | 2 Months
To evaluate the reliability of different skin elasticity measurement on the cheek between different time points and different technicians. | 2 Months
To evaluate the reliability of spectrophotometric skin color measurement on the cheek between different time points and different technicians. | 2 Months
To evaluate the reliability of epidermal thickness measurement on the cheek between different time points and different technicians. | 2 Months
To evaluate the reliability of different skin probe measurements and imaging modalities on changes in skin roughness on the cheek between different time points and different technicians. | 2 Months
To evaluate the reliability of different skin probe measurements and imaging modalities on changes in skin gloss on the cheek between different time points and different technicians. | 2 Months
To evaluate the reliability of skin gloss measurement on the cheek between different technicians. | 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Siham Rharbaoui, MD, Principal Investigator — DERMSCAN - Pharmascan
Locations (1):
- Dermscan-Pharmascan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance — http://www.allerganclinicaltrials.com/